CLINICAL TRIAL: NCT05863325
Title: An Open-label, Randomized, Positive Drug-controlled Phase Ⅱ Study to Compare the Efficacy and Safety of HB1801 to Taxotere in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Compare the Efficacy and Safety of HB1801 to Taxotere in Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-009
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Locally Advanced or Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB1801 (Experimental): HB1801 will be given in 21-day cycles until documented disease progression, discontinuation due to toxicity, withdrawal of consent, initiation of a new antitumor therapy, loss of follow-up, death, or study completion, whichever occurs first.
  Interventions: Drug: HB1801
- Taxotere (Active Comparator): Taxotere will be given in 21-day cycles until documented disease progression, discontinuation due to toxicity, withdrawal of consent, initiation of a new antitumor therapy, loss of follow-up, death, or study completion, whichever occurs first.
  Interventions: Drug: Taxotere

INTERVENTIONS:
Drug: HB1801 — HB1801 will be administered by intravenous (IV) injections on the first day of each cycle.
  Arms: HB1801
Drug: Taxotere — Taxotere will be administered by intravenous (IV) injections on the first day of each cycle.
  Arms: Taxotere

SUMMARY:
This is an open-label, randomized, positive drug-controlled Phase Ⅱ clinical study to compare the efficacy and safety of HB1801 to Taxotere in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who have failed platinum- containing chemotherapies.

DETAILED DESCRIPTION:
Eligible patients will enter the screening period up to 28 days before the start of treatment. Patients will be randomized in a 1:1 ratio to receive HB1801 (trial group) or Taxotere (control group). Randomized stratification factor is pathological type (squamous vs. non-squamous). Patients in trial group will receive HB 1801 and patients in control group will receive Taxotere. HB 1801 or Taxotere will be given on the first day of each cycle (21 days). Each patient will be treated until documented disease progression, discontinuation due to toxicity, withdrawal of consent, initiation of a new antitumor therapy, loss of follow-up, death, or study completion, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. Voluntarily signed written informed consent form, willing and able to comply with scheduled visits and treatment and laboratory tests of the protocol.
3. Patient has a diagnosis of locally advanced or metastatic NSCLC as determined by histological or cytological results.
4. Patients with known EGFR-sensitive mutation /ALK fusion /ROS1 fusion must have been documented disease progression during or after targeted drugs treatments and platinum-containing chemotherapies; Patients without above positive genes must have been documented disease progression during or after PD-1/PD-L1 inhibitors treatments and platinum-containing chemotherapies (combined or sequential). Note: For prior adjuvant/neoadjuvant treatment with platinum-containing regimens of chemotherapy, progression during or within 6 months of completion of adjuvant/neoadjuvant treatment may be considered a failure of platinum-containing chemotherapy.
5. At least one measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
6. Adequate organ function.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Patients of reproductive potential must be willing to use adequate contraception during the study and through 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Prior use of docetaxel monotherapy or combination therapy for metastatic disease.
2. Known ≥ grade 3 hypersensitivity and/or contraindications to human albumin or docetaxel; known allergy and/or contraindications to glucocorticoids (including but not limited to active digestive tract ulcers, severe hypertension, severe hypokalemia, glaucoma, etc.).
3. Leptomeningeal metastases and/or untreated active brain metastases; if the patient's brain metastases have been treated, a stable state is required prior to randomization (no radiographically confirmed progression and normal return of all neurologically relevant symptoms within 4 weeks prior to randomization), no new brain metastases or enlargement of the original brain metastases are shown on radiographs, and steroid hormone therapy is not required for at least 7 days prior to randomization.
4. History of other malignancies within 3 years prior to randomization, excluding basal cell or squamous cell carcinoma of skin and cervical carcinoma in situ that have been radically treated.
5. Serosal effusion requiring drainage or diuretic treatment (such as pleural effusion, peritoneal effusion, or pericardial effusion) within 2 weeks before randomization.
6. History of severe cardiovascular disease within 6 months prior to randomization, including but not limited to:

（1) Uncontrolled hypertension (defined as persistent systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg despite the use of antihypertensive medications); （2) Severe arrhythmias and conduction abnormalities requiring treatment with antiarrhythmic agents other than beta-blockers or digoxin (except atrial fibrillation and paroxysmal supraventricular tachycardia); （3) History of myocardial infarction, unstable angina pectoris, angioplasty, and coronary artery bridging surgery; （4) Heart failure, New York Heart Association (NYHA)≥grade 3; （5) QTcF > 480 ms; （6) Other heart diseases that investigators identify as clinically significant. 7. Active infection treated with intravenous antibiotics within 2 weeks prior to randomization.

8. Patients who have undergone major organ surgery (excluding needle biopsy) within 4 weeks prior to randomization or who will require elective surgery during the trial period.

9. The toxicity of previous anti-tumor therapy does not return to grade≤1 (CTCAE v5.0), except for grade 2 neuropathy, alopecia, hypothyroidism caused by prior anti-tumor therapy (including hormone replacement therapy), and toxicity judged by the investigator to be of no safety risk.

10. Receiving antitumor therapy such as chemotherapy, targeted therapy, immunotherapy, and other investigational agents within 4 weeks or 5 half-lives (whichever is shorter but at least 2 weeks) prior to randomization, other conditions as follows: Received radiotherapy within 2 weeks prior to randomization, or received radiotherapy prior to 2 weeks of randomization but patient has not recovered from all acute toxicity and requires hormone therapy; Chinese medicines with anti-tumor indications administered within 2 weeks prior to randomization.

11. Use of potent inhibitors or potent inducers of CYP3A4 within 2 weeks prior to randomization.

12. Life expectancy < 3 months. 13. HBsAg/HBcAb positive with HBV-DNA ≥ 10^2 cps/mL or ≥ 2000 IU/mL); hepatitis C antibody-positive with a positive PCR result for HCV RNA; Patients infected with human immunodeficiency virus (HIV); Patients with active tuberculosis.

14. Patients are not suitable for the study in the investigator's opinion, include but are not limited to, conditions in which the patient has a serious or uncontrolled medical condition, interferes with the interpretation of the study results, and interferes with compliance with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to approximately 3 years

SECONDARY OUTCOMES:
Progression-free Survival（PFS） | up to approximately 3 years
Disease Control Rate（DCR） | up to approximately 3 years
Duration of Response (DoR) | up to approximately 3 years
Overall Survival (OS) | up to approximately 3 years
Frequency and Severity of Adverse Events During Treatment | up to approximately 3 years
Total and Free Docetaxel Concentrations in Plasma | The first cycle (21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Provincial Tumor Hospital, Changchun, Jilin, China